CLINICAL TRIAL: NCT01386957
Title: Steroid Treatment of Childhood Idiopathic Nephrotic Syndrome: Epidemiology, Therapeutic Adequacy, Medium and Long Term Outcomes. A Prospective Observational Cohort Study.
Brief Title: Steroid Treatment of Idiopathic Nephrotic Syndrome
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: IL Sogno di Stefano (Other); Nando and Elsa Peretti Foundation (Other)
Responsible Party: Principal Investigator, Giovanni Montini, MD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: SNI-NET 2011
Record Dates: First submitted 2011-06-30; First posted 2011-07-01 (Estimated); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Nephrotic Syndrome
Keywords: Nephrotic Syndrome; Steroid treatment; Proteinuria; Child
MeSH Terms: conditions — Nephrotic Syndrome; Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole Blood and Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: children aged 6 months - 18 years, diagnosed with an initial episode of INS occurring from the first of July 2011 to the 31st of june 2013.

SUMMARY:
Idiopathic nephrotic syndrome (INS) is the most frequent glomerular disease in childhood. Currently, all children with INS are treated at onset with steroids. The optimal duration and dosage of steroid therapy is debated. For each patient, the challenge is to minimise potential side effects of steroids, while achieving a good clinical response.

The aim of our study is to assess the benefits and potential adverse effects of a prolonged initial corticosteroid regimen, for the treatment of the initial episode. The results will be compared with data obtained retrospectively. In addition genetic studies will be undertaken with the aim of evaluating pharmacodynamics of steroid treatment with the ultimate goal to individualise treatment in single patients.

1. Study group: children aged 6 months - 18 years, diagnosed with an initial episode of idiopathic nephrotic syndrome
2. Control group: data of children with a onset INS between January 2007 and December 2009 from the same area of the study group and treated with a short steroid regimen will be retrospectively analysed and compared

DETAILED DESCRIPTION:
Background Idiopathic nephrotic syndrome (INS) is the most frequent glomerular disease in childhood, with an incidence of 2-4 cases per 100,000 children. Currently, all children with INS are treated at onset with steroids. Approximately 80% of cases respond to oral corticosteroid therapy, but 75-80% of these children will experience relapses which can recur over many years. The optimal duration and dosage of steroid therapy at onset and during subsequent relapses is debated. For each patient, the challenge is to minimise potential side effects of steroid therapy (hypertension, bone disease, Cushing syndrome, obesity, growth retardation, cataracts and a variety of psychological, social and behavioural disturbances) while achieving a good clinical response. This is particularly difficult at the beginning of the illness, because of the lack of reliable indicators that allow the identification of patients who will respond poorly or will experience frequent relapses. In 2006 the Cochrane Collaboration published the first systematic review of corticosteroid therapy for childhood idiopathic nephrotic syndrome. They concluded that children with the first episode of steroid sensitive INS should be treated for a minimum of three months, to achieve a reduction in the subsequent relapse rate.

The fine border between the optimal dose of steroids and the collateral effects can not be overlooked given the results of some recent studies (relative to patients with chronic inflammatory bowel disease or children with acute lymphoblastic leukemia subject to prolonged cycles of steroid therapy) based on the pharmacogenetic evaluation of the diverse individual responses to steroids. Clinical data supports the concept that the collateral effects of steroids are not exclusively dose related, but can depend on constitutional hypersensitivity or resistance, at times specific for a particular corticosteroid.

This diverse individual response can depend on a number of factors. The activity of the corticosteroids is mediated by interactions with the DNA (genomic mechanism) or by a direct interaction with the cellular membranes (non-genomic mechanism). The genomic effects are by far the most important and are mediated by the interactions of the steroids with a specific cytoplasmic receptor (GR). The binding of the steroid determines the activation of the receptor and its translocation within the nucleus where it induces (transactivation) or inhibits (transcriptional interference) the synthesis of numerous regulatory proteins. The mechanism of transactivation is likely responsible for the major part of collateral effects (suppression of the hypothalamic-hypophysial-adrenal axis, genesis of glaucoma and diabetes), while the anti-inflammatory effects are for the most part tied to transcriptional inhibition (with reduced synthesis of pro-inflammatory cytokines, cyclic oxygenase2, inducible forms of nitrite synthesis and finally a reduction in synthesis of receptors for Fc and C3).

There are individual diverse molecular anomalies of the gene for the glucocorticoid receptors (hGR/NR3C1) that have bean uncovered: for example the presence of polymorphisms of the gene hGR is correlated with receptor hyperactivity (Bcl1 e N3635) or relative resistance of the glucocorticoid receptor (polymorphism ER22/23EK); a further 15 mutations have already been identified to be associated with corticosteroid resistance.

These facts open interesting possibilities for pharmacological research with the hypothesis of being able to adjust steroid therapy in response to an individuals genetic make-up and predict the appearance of side effects.

AIM The aim of our study is to assess the benefits and potential adverse effects of a prolonged initial corticosteroid regimen across four Italian regions, for the treatment of the initial episode of INS. The results will be compared with data obtained retrospectively from the analysis of a control group of INS, treated with a short steroid regimen during the previous 3 years in the same area. In addition genetic studies will be undertaken with the aim of evaluating pharmacogenetics and pharmacodynamics of steroid treatment with the ultimate goal to individualise treatment in single patients.

Study population:

1. Study group: children aged 6 months - 18 years, diagnosed with an initial episode of idiopathic nephrotic syndrome (proteinuria> 40mg/m2/h or urine protein/creatine ratio > 2 mg/mg and hypoalbuminemia <2.5g/dL).

   Subjects will be enrolled from the first of July 2011 to the 30th of June 2013; the follow-up of each subject will continue for 24 months.
2. Control group: data of children with a onset INS between January 2007 and December 2009 from the same area of the study group and treated with a short steroid regimen will be retrospectively analysed and compared. Data will be recorded anonymously through an online database. The epidemiological, clinical, therapeutic parameters collected will be the same of the intervention group, except for pharmacogenetic and pharmacodynamic tests, and behavioral questionnaires.

All study group patients will be subjected to the following protocol:

Induction therapy: prednisone 60mg/m2/day in 2 divided doses. Patients achieving remission within 10 days, will continue this dosage until the 28th day, whereas patients not achieving remission within 10 days, will continue this dosage until the 42nd day. Moreover, from the 3rd day of remission prednisone will be given in a single morning dose.

Maintenance therapy:

Patients going into remission during the induction therapy will have steroids tapered over a 16 weeks period:

* 40 mg/m2/alt day in a single morning dose for 4 weeks,
* 30 mg/m2/alt day in a single morning dose for 2 weeks,
* 22.5 mg/m2/alt day in a single morning dose for 2 weeks,
* 15 mg/m2/alt day in a single morning dose for 2 weeks,
* 7.5 mg/m2/alt day in a single morning dose for 2 weeks,
* 4.5 mg/m2/alt day in a single morning dose for 4 weeks,
* stop therapy. A subgroup of patients (estimated to be 100) will undergo pharmacogenetic and pharmacodynamic studies. The pharmacogenetic study will evaluate the presence of gene polymorphisms that modifies the numbers of functioning receptors and their affinity for steroids (genes studied are showed in Tab 3). The pharmacodynamic study will evaluate the in vitro response to steroids on blood mononuclear cells: individual sensibility to steroids will be detected before and during steroid treatment and compared with the clinical response, in order to tailor treatment in the future.

Relapses. Relapses will be treated with a further prolonged steroid regimen witch is described in the protocol per extenso.

Patient monitoring:

1. Clinical examination Height, weight, BMI, blood pressure Parent heights recording (for familial target) (at onset, remission, 4th, 20th weeks, 6, 12, 18, 24 months)
2. Biochemistry (at onset, 4th week, 24 months)

   Blood CBC; serum glycemia, urea, creatinine, uric acid, proteins, albumin, cholesterol, HDL, LDL, triglycerides, a2globulins, gammaglobulins, PT, PTT, fibrinogen, Anti-Thrombin III°, Na, K, Cl, Ca, P, blood sample for pharmacogenetic and pharmacodynamic study

   Urine Urine examination. Proteinuria and creatininuria on a 24h sample
3. Behavioral questionnaires(at onset, 4th, 6, 12, 24 months)

ASEBA CBCL Achenbach System of Empirically Based Assessment Child Behavior Checklist.

EQ-5D-PROXY EuroQol Group (version for parents) PedsQL Pediatric Quality of Life Inventory (version for parents and children) EQ-5D-Y EuroQol Group (version for children)

The following epidemiological and therapeutical data will be collected

Epidemiological data

* Sex
* Age at onset
* Season
* Ethnicity
* Days of hospitalization.
* Number of blood tests performed during the follow-up

Therapeutic data

* Time to remission (days), number of relapses at 6-12-24 months
* Time and total dose (mg/m2) of induction therapy
* Time and total dose (mg/m2) of maintenance therapy
* Prednisone total dose at the end of the 2yrs of follow-up
* Albumin infusions (g/kg/patient)
* Use of albumin infusions and diuretics
* Number of immunosuppressive drugs associated to prednisone (and total dose in mg/kg)

ELIGIBILITY:
Inclusion Criteria:

1. Age > 6 months and< 18 years
2. Idiopathic nephrotic syndrome
3. Ethical committee approval

Exclusion Criteria:

1. Age < 6 months or > 18 years
2. Congenital nephrotic syndrome
3. Secondary nephrotic syndrome (post-infectious, SLE, Schonlein-Henoch) defined by clinical features, low C3 and C4 levels, severe hypertension and macrohematuria
4. nephrotic syndrome associated to other syndromes (Dennys Drash, Frasier syndrome, et.cet) or to Wilms'tumor.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 6 months - 18 years, diagnosed with an initial episode of idiopathic nephrotic syndrome (proteinuria> 40mg/m2/h or urine protein/creatine ratio > 2 mg/mg and hypoalbuminemia <2.5g/dL).
  Subjects will be enrolled from the first of July 2011 to the 31st of June 2013 from the following Italian regions Emilia Romagna, Lombardia, Toscana, Trentino Alto Adige, Friuli Venezia Giulia, Marche and Sicilia; the follow-up of each subject will continue for 24 months.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2011-07; Primary Completion 2016-11 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Montini, MD, Study Chair — Azienda Ospedaliero-Universitaria Sant'Orsola Malpighi, Bologna, Italy
Locations (11):
- Italy (11):
  - Azienda Ospedaliera-Universitaria Sant'Orsola Malpighi, Bologna, Emilia-Romagna
  - PO Salesi, SOS Centro di Riferimento Regionale di Nefrologia e Dialisi Pediatrica, Ancona
  - Ospedale Pediatrico Giovanni XXIII, Bari
  - Azienda Ospedaliera Universitaria Meyer, SOD Complessa Nefrologia Pediatrica, Florence
  - Istituto Giannina Gaslini, Dept of Pediatric Nephrology, Genova
  - AOU Policlinico G Martino UOS dipartimentale Nefrologia e Reumatologia pediatrica, Messina
  - Fondazione IRCCS Ca' Granda Ospedale MAggiore Policlinico, UOC Nefrologia e Dialisi, Milan
  - Ospedale dei bambini Di Cristina, UOC Nefrologia Pediatrica, Palermo
  - Ospedale degli Angeli, Dept of Pediatrics, Pordenone
  - Ospedale Pediatrico Burlo Garofalo, Trieste
  - Università di Trieste, Department of Life Sciences, Trieste

REFERENCES:
- [Derived] Nardini B, La Scola C, Corrado C, Edefonti A, Giordano M, Pillon R, Mastrangelo AP, Materassi M, Alberici I, Morello W, Puccio G, Montini G, Pasini A. Time to remission in childhood steroid sensitive nephrotic syndrome: a change in perspective. Eur J Pediatr. 2025 Mar 20;184(4):262. doi: 10.1007/s00431-025-06090-z. PMID 40111516
- [Derived] Pasini A, Bertulli C, Casadio L, Corrado C, Edefonti A, Ghiggeri G, Ghio L, Giordano M, La Scola C, Malaventura C, Maringhini S, Mastrangelo AP, Materassi M, Mencarelli F, Messina G, Monti E, Morello W, Puccio G, Romagnani P, Montini G; NefroKid Study Group. Childhood Idiopathic Nephrotic Syndrome: Does the Initial Steroid Treatment Modify the Outcome? A Multicentre, Prospective Cohort Study. Front Pediatr. 2021 Jul 8;9:627636. doi: 10.3389/fped.2021.627636. eCollection 2021. PMID 34307246
- [Derived] Pasini A, Aceto G, Ammenti A, Ardissino G, Azzolina V, Bettinelli A, Cama E, Cantatore S, Crisafi A, Conti G, D'Agostino M, Dozza A, Edefonti A, Fede C, Groppali E, Gualeni C, Lavacchini A, Lepore M, Maringhini S, Mariotti P, Materassi M, Mencarelli F, Messina G, Negri A, Piepoli M, Ravaglia F, Simoni A, Spagnoletta L, Montini G; NefroKid Study Group. Best practice guidelines for idiopathic nephrotic syndrome: recommendations versus reality. Pediatr Nephrol. 2015 Jan;30(1):91-101. doi: 10.1007/s00467-014-2903-7. Epub 2014 Aug 17. PMID 25127916